CLINICAL TRIAL: NCT02058693
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study of Adjunctive, Flexible-Dose Mixed Salts Amphetamine in Adult Outpatients With Major Depressive Disorder (MDD) Responding Inadequately to Current Antidepressant Therapy
Brief Title: Adjunctive Mixed Salts Amphetamine for Depressed Adults With Incomplete Response to Current Antidepressant Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTHF-1
Record Dates: First submitted 2014-01-15; First posted 2014-02-10 (Estimated); Results first posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Adderall

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1(A): Placebo/MSA (Placebo Comparator): Phase I (3 weeks) placebo adjunctive to Anti-Depressant Therapy (ADT). The total daily dosing of the concurrent ADT will be as follow: escitalopram 10-40 mg; Fluoxetine 20-80 mg; paroxetine controlled release (CR) 25-100 mg (paroxetine 20-80 mg may be substituted if paroxetine CR is not available); sertraline 100-400 mg; venlafaxine extended release (XR) 150-600 mg; desvenlafaxine 50-200 mg; citalopram 20-80 mg; or duloxetine 60-180 mg; buproprion 150-450 mg; mirtazapine 15-45 mg, tricyclics (standard dosing, individually per label instructions).
  Phase II (3 weeks) mixed salts amphetamine adjunctive to ADT (as in Phase I).
  Interventions: Drug: mixed salts amphetamine
- Group 2(B): MSA/MSA (Active Comparator): Phase I (3 weeks) mixed salts amphetamine adjunctive to Anti-Depressant Therapy (ADT). The total daily dosing of the concurrent ADT will be as follow: escitalopram 10-40 mg; Fluoxetine 20-80 mg; paroxetine controlled release (CR) 25-100 mg (paroxetine 20-80 mg may be substituted if paroxetine CR is not available); sertraline 100-400 mg; venlafaxine extended release (XR) 150-600 mg; desvenlafaxine 50-200 mg; citalopram 20-80 mg; or duloxetine 60-180 mg; buproprion 150-450 mg; mirtazapine 15-45 mg, tricyclics (standard dosing, individually per label instructions).
  Phase II (3 weeks) mixed salts amphetamine adjunctive to ADT (as in Phase I).
  Interventions: Drug: mixed salts amphetamine

INTERVENTIONS:
Drug: mixed salts amphetamine — adjunctive to ADT
  Other Names: Adderall

SUMMARY:
In this Phase 4 trial we will study the safety, tolerability and efficacy of mixed salts amphetamine (MSA), trade name Adderall, augmentation of antidepressant therapy for Major Depressive Disorder (MDD) in depressed outpatient adults who are taking an antidepressant but have not had complete resolution of their symptoms.

DETAILED DESCRIPTION:
Forty adult outpatients with MDD who failed at least one adequate trial of antidepressant monotherapy will be consented in a 63-day, cross-sequential, multicenter study comprising two treatment phases of 21 days each. The time frame from consent to baseline is 7 days. Patients will receive placebo or MSA in Phase 1, and in Phase 2, participants will receive MSA. There will also be a two-week follow up visit after the completion of Phase 2.

We hypothesize that MSA will be safe and well tolerated, and will improve the patient's response to their antidepressant and provide superior symptom relief to antidepressant alone. The primary outcome measure is the Massachusetts General Hospital Cognitive-Physical Function Questionnaire (MGH-CPFQ).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female outpatients between the ages of 18-70.
2. Subject must meet criteria for single or recurrent, non-psychotic episode of MDD according to Diagnostic and Statistical Manual IV Text Revised (DSM-IV-TR) diagnosis, as determined by Structured Clinical Inventory of Depressive Symptoms (SCID) and confirmed by assessment of investigator.
3. Current depressive episode must be at least 8 weeks in duration.
4. Hamilton Depression Rating Scale 17 (HDRS-17) score ≥ 14 at both the screen and baseline visits.
5. Subject must have been receiving an adequate, stable dose of ADT, based on Massachusetts General Hospital-Antidepressant Treatment Response Questionnaire (MGH-ATRQ).
6. Subject must be responding inadequately to his/her current monotherapy ADT in the current major depressive episode (MDE).
7. Subjects must be able to read and understand English and be able to provide written informed consent.
8. Subjects must be considered reliable, able to comply with protocol requirements and understand the risks and benefits, per the investigator's clinical judgment.
9. Female subjects of childbearing potential must agree to use adequate form of birth control throughout the course of the study.

   -

Exclusion Criteria:

1. Inadequate response during the current episode to more than 3 adequate trials of an ADT, as defined by the MGH-ATRQ.
2. Psychiatric hospitalization within the last 6 months.
3. Presence of cognitive disorder(s), bipolar disorder, Axis II pathology or other condition that investigator believes would interfere with participation in the study.
4. Substance use disorder, current (as defined by DSM-IV-TR SCID) or positive results on urine drug screen or laboratory blood tests.
5. Risk to self or others.
6. The presence of any medical condition, current or past, stable or unstable, that contraindicates the use of antidepressant medication or mixed amphetamine salts medication as determined by clinician's judgment.
7. Clinically significant abnormal findings on physical exam, EKG or laboratory tests; current unstable, untreated hypertension in the opinion of the investigator; history of cerebrovascular accident (CVA) or seizure disorder (other than febrile childhood seizure).
8. Allergies and/or adverse drug reactions to MSA.
9. Failure to respond to an adequate trial of MSA adjunctive to ADT in the current episode.
10. Subjects taking narcotics, herbal/homeopathic remedies and/or other substance with psychotropic activity, based upon clinical judgment of study investigator.
11. Pregnant or breastfeeding women.

    -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2010-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corey N Goldstein, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1(A): Placebo/MSA: Phase I (3 weeks) placebo adjunctive to Anti-Depressant Therapy (ADT). The total daily dosing of the concurrent ADT will be as follow: escitalopram 10-40 mg; Fluoxetine 20-80 mg; paroxetine CR (controlled release) 25-100 mg (paroxetine 20-80 mg may be substituted if paroxetine CR is not available); sertraline 100-400 mg; venlafaxine XR (extended release) 150-600 mg; desvenlafaxine 50-200 mg; citalopram 20-80 mg; or duloxetine 60-180 mg; buproprion 150-450 mg; mirtazapine 15-45 mg, tricyclics (standard dosing, individually per label instructions).
  Phase II (3 weeks) mixed salts amphetamine adjunctive to ADT
- Group 2(B): MSA/MSA: Phase I (3 weeks): mixed salts amphetamine, adjunctive to Anti-Depressant Therapy (ADT). The total daily dosing of the concurrent ADT will be as follow: escitalopram 10-40 mg; Fluoxetine 20-80 mg; paroxetine CR (controlled release) 25-100 mg (paroxetine 20-80 mg may be substituted if paroxetine CR is not available); sertraline 100-400 mg; venlafaxine XR (extended release) 150-600 mg; desvenlafaxine 50-200 mg; citalopram 20-80 mg; or duloxetine 60-180 mg; buproprion 150-450 mg; mirtazapine 15-45 mg, tricyclics (standard dosing, individually per label instructions).
  Phase II (3 weeks) mixed salts amphetamine adjunctive to ADT
Period: Phase 1
Arm/Group | Group 1(A): Placebo/MSA | Group 2(B): MSA/MSA
Started | 21 | 20
Completed | 16 | 16
Not Completed | 5 | 4
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Physician Decision | 1 | 1
Period: Phase 2
Arm/Group | Group 1(A): Placebo/MSA | Group 2(B): MSA/MSA
Started | 16 | 16
Completed | 16 | 14
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Group 1(A): Placebo/MSA: Phase I (3 weeks) placebo adjunctive to Anti-Depressant Therapy (ADT). The total daily dosing of the concurrent ADT will be as follow: escitalopram 10-40 mg; Fluoxetine 20-80 mg; paroxetine CR (controlled release) 25-100 mg (paroxetine 20-80 mg may be substituted if paroxetine CR is not available); sertraline 100-400 mg; venlafaxine XR (extended release) 150-600 mg; desvenlafaxine 50-200 mg; citalopram 20-80 mg; or duloxetine 60-180 mg; buproprion 150-450 mg; mirtazapine 15-45 mg, tricyclics (standard dosing, individually per label instructions).
  Phase II (3 weeks) mixed salts amphetamine adjunctive to ADT
  mixed salts amphetamine: adjunctive to ADT
- Group 2(B): MSA/MSA: mixed salts amphetamine, adjunctive to Anti-Depressant Therapy (ADT). The total daily dosing of the concurrent ADT will be as follow: escitalopram 10-40 mg; Fluoxetine 20-80 mg; paroxetine CR (controlled release) 25-100 mg (paroxetine 20-80 mg may be substituted if paroxetine CR is not available); sertraline 100-400 mg; venlafaxine XR (extended release) 150-600 mg; desvenlafaxine 50-200 mg; citalopram 20-80 mg; or duloxetine 60-180 mg; buproprion 150-450 mg; mirtazapine 15-45 mg, tricyclics (standard dosing, individually per label instructions).
  Phase II (3 weeks) mixed salts amphetamine adjunctive to ADT
  mixed salts amphetamine: adjunctive to ADT
- Total: Total of all reporting groups
Arm/Group | Group 1(A): Placebo/MSA | Group 2(B): MSA/MSA | Total
Number analyzed (Participants) | 21 | 20 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 19 | 40
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 24
  Male | 8 | 9 | 17
Region of Enrollment [Number; unit: participants]
  United States | 21 | 20 | 41

OUTCOME MEASURES:

1. Primary Outcome: Change in Scores on the Massachusetts General Hospital Cognitive and Physical Functioning Questionnaire (MGH-CPFQ)
Description: The CPFQ is a seven-item self-administered questionnaire with higher scores indicating increased impairment in cognitive and physical functioning; score range being 7-42.
Time Frame: Baseline (Visit 2); End Phase I (Visit 5, Week 3): End Phase II (Visit 8, Week 6)
Population: Subjects completing all seven visits and administered the CPFQ. Some subjects completing seven visits were not administered the CPFQ in error.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Group 1(A): Placebo/MSA | Group 2(B): MSA/MSA
Number analyzed (Participants) | 10 | 13
Scores on a scale
  Baseline (V2) | 27.5 (8.4896) | 29 (5.33)
  End Phase I (V5; W3) | 22.6 (7.78) | 25 (6.45)
  End Phase II (V8; W6) | 16 (4.69) | 21 (5.73)

2. Secondary Outcome: Change in Scores of the Montgomery Asberg Depression Rating Scale (MADRS)
Description: The group treated with mixed salt amphetamine (MSA) adjunctive to antidepressant therapy (ADT) will show a greater mean change from baseline to endpoint as compared to the group treated with placebo (PBO) adjunctive to ADT as measure by the change ion the MADRS scores.
  The MADRS is clinician-rated and consists of 10 items; each item is rated on a 0-6 scale, resulting in a maximum total score of 60 points, with higher scores indicative of greater depressive symptomology. The MADRS scoring instructions indicate that a total score ranging from 0 to 6 indicates that the patient is in the normal range (no depression), a score ranging from 7 to 19 indicates "mild depression," 20 to 34 indicates "moderate depression," a score of 35 and greater indicates "severe depression." There is evidence that an improvement of two points or more on the MADRS is considered clinically relevant.
Time Frame: Baseline (Visit 2); End Phase I (Visit 5, Week 3): End Phase II (Visit 8, Week 6)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Group 1(A): Placebo/MSA: Phase I (3 weeks) placebo adjunctive to Anti-Depressant Therapy (ADT). The total daily dosing of the concurrent ADT will be as follow: escitalopram 10-40 mg; Fluoxetine 20-80 mg; paroxetine controlled release (CR) 25-100 mg (paroxetine 20-80 mg may be substituted if paroxetine CR is not available); sertraline 100-400 mg; venlafaxine extended release (XR) 150-600 mg; desvenlafaxine 50-200 mg; citalopram 20-80 mg; or duloxetine 60-180 mg; buproprion 150-450 mg; mirtazapine 15-45 mg, tricyclics (standard dosing, individually per label instructions).
  Phase II (3 weeks) mixed salts amphetamine adjunctive to ADT (as in Phase I).
  mixed salts amphetamine: adjunctive to ADT
- Group 2(B): MSA/MSA: Phase I (3 weeks) mixed salts amphetamine adjunctive to Anti-Depressant Therapy (ADT). The total daily dosing of the concurrent ADT will be as follow: escitalopram 10-40 mg; Fluoxetine 20-80 mg; paroxetine controlled release (CR) 25-100 mg (paroxetine 20-80 mg may be substituted if paroxetine CR is not available); sertraline 100-400 mg; venlafaxine extended release (XR) 150-600 mg; desvenlafaxine 50-200 mg; citalopram 20-80 mg; or duloxetine 60-180 mg; buproprion 150-450 mg; mirtazapine 15-45 mg, tricyclics (standard dosing, individually per label instructions).
  Phase II (3 weeks) mixed salts amphetamine adjunctive to ADT (as in Phase I).
  mixed salts amphetamine: adjunctive to ADT
Arm/Group | Group 1(A): Placebo/MSA | Group 2(B): MSA/MSA
Number analyzed (Participants) | 11 | 13
Scores on a scale
  Baseline (V2) | 24.18 (6.54) | 27 (6.2)
  End of Phase I (V5; W3) | 11.55 (7.67) | 18.31 (10.24)
  End of Phase II (V8; W6) | 7.10 (4.76) | 10.17 (8.33)

3. Secondary Outcome: Change in Scores on the Quick Inventory of Depressive Symptomatology Self Report 16 (QIDS-SR-16)
Description: The group with mixed salt amphetamine (MSA) adjunctive to antidepressant therapy (ADT) will show statistically significant improvement in core residual symptoms of major depressive disorder (MDD) extant on monotherapy ADT as measured by the Quick Inventory of Depressive Symptomatology Self Report 16.
  16 items comprising 9 domains; each domain is scored from 0 to 3, with higher scores reflecting greater psychopathology. Total scores range from 0 to 27. Scoring procedure is to include ONLY the highest score on among the 4 sleep items (items 1 to 4); include ONLY the highest score among the 4 weight items (items 6 to 9); include ONLY the highest score on either of the 2 psychomotor items (15 and 16). The scores for these 3 domains are then added to the scores (0-3) for each of the 6 MDD symptom domains for a total score of 0-27.
Time Frame: Baseline (Visit 2); End Phase I (Visit 5, Week 3): End Phase II (Visit 8, Week 6)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Group 1(A): Placebo/MSA | Group 2(B): MSA/MSA
Number analyzed (Participants) | 11 | 13
Scores on a scale
  Baseline (V2; W1) | 12.5 (3.8) | 14 (4.5)
  End of Phase I (V5; W3) | 7.8 (3.22) | 8.7 (5.6)
  End of Phase II (V7; W6) | 5 (2.2) | 5.3 (4.4)

ADVERSE EVENTS:
Time Frame: AE data were collected over the seven weeks of the trial.
Description: Definition does not differ from the clinicaltrials.gov definitions. Adverse event data were collected by group but not by phase in this trial.
Groups:
- Group 1(A): Placebo/MSA: Phase I (3 weeks) placebo adjunctive to Anti-Depressant Therapy (ADT). The total daily dosing of the concurrent ADT will be as follow: escitalopram 10-40 mg; Fluoxetine 20-80 mg; paroxetine CR (controlled release) 25-100 mg (paroxetine 20-80 mg may be substituted if paroxetine CR is not available); sertraline 100-400 mg; venlafaxine XR (extended release) 150-600 mg; desvenlafaxine 50-200 mg; citalopram 20-80 mg; or duloxetine 60-180 mg; buproprion 150-450 mg; mirtazapine 15-45 mg, tricyclics (standard dosing, individually per label instructions).
  Phase II (3 weeks) mixed salts amphetamine adjunctive to ADT (as in Phase I).
  mixed salts amphetamine: adjunctive to ADT
- Group 2(B): MSA/MSA: Phase I (3 weeks) mixed salts amphetamine adjunctive to Anti-Depressant Therapy (ADT). The total daily dosing of the concurrent ADT will be as follow: escitalopram 10-40 mg; Fluoxetine 20-80 mg; paroxetine CR (controlled release) 25-100 mg (paroxetine 20-80 mg may be substituted if paroxetine CR is not available); sertraline 100-400 mg; venlafaxine XR (extended release) 150-600 mg; desvenlafaxine 50-200 mg; citalopram 20-80 mg; or duloxetine 60-180 mg; buproprion 150-450 mg; mirtazapine 15-45 mg, tricyclics (standard dosing, individually per label instructions).
  Phase II (3 weeks) mixed salts amphetamine adjunctive to ADT (as in Phase I).
  mixed salts amphetamine: adjunctive to ADT
Arm/Group | Group 1(A): Placebo/MSA | Group 2(B): MSA/MSA
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 8/16 | 9/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1(A): Placebo/MSA (N=16) | Group 2(B): MSA/MSA (N=16)
Agitation (Nervous system disorders) | 2 (2) | 2 (2) — Reported subjective experience of feeling "jittery," edgy," or "muscle tension."
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Bad taste (Product Issues) | 1 (1) | 0 (0)
Blurred vision (General disorders) | 1 (1) | 0 (0)
Body ache (General disorders) | 1 (1) | 1 (1) — Any reported bodily aches
Bruising (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
Decreased appetite (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry mouth (General disorders) | 1 (1) | 2 (2)
Headache (General disorders) | 4 (4) | 4 (4)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Insomnia (General disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Mild heart tremor (Cardiac disorders) | 1 (1) | 1 (1)
Racy feelings (Psychiatric disorders) | 0 (0) | 1 (1)
Acid reflux (Gastrointestinal disorders) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Injury: slip and fall, bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sweating (General disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Tinnitus (General disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Vertigo (General disorders) | 1 (1) | 0 (0)
Watery, itchy eyes (Immune system disorders) | 1 (1) | 0 (0)
Weight loss (General disorders) | 0 (0) | 1 (1)
Word finding (Psychiatric disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2013-09-25): https://cdn.clinicaltrials.gov/large-docs/93/NCT02058693/Prot_SAP_000.pdf
  • Informed Consent Form (2013-09-25): https://cdn.clinicaltrials.gov/large-docs/93/NCT02058693/ICF_001.pdf